CLINICAL TRIAL: NCT02369094
Title: A Study on Effects of Acupressure Among the Frail Elderly in the Social Centers for the Elderly and Neighbourhood Elderly Centers of Yan Chai Hospital, Social Services Department (YCHSS)
Brief Title: A Study on Effects of Acupressure Among the Frail Elderly in the Community Dwellings
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Collaborators: Yan Chai Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CTC1215
Record Dates: First submitted 2015-02-04; First posted 2015-02-23 (Estimated); Last update posted 2016-07-14 (Estimated); Status verified 2016-07

CONDITIONS: Impaired
Keywords: Frailty; Frail elderly; Acupressure; Pragmatic Randomised Controlled Trial
MeSH Terms: conditions — Frailty | interventions — Acupressure

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Acupressure Group (Experimental): A 15 minutes structured acupressure protocol with specific acupoints and applications technique will be performed on the elderly participants twice a week by the research team in YCHSS centers. The caregiver of the elderly will be trained and perform the same acupressure protocol on the elderly at 2 additional occasions during the week. The total trial period is 12 weeks.
  Interventions: Other: acupressure
- Waiting Control Group (Other): No acupressure therapy will be provided during the 1st 12 weeks' of study.The enrolled elderly will join a group activity, resembling the other group activities that held in that particular center, their caregivers will be requested to spend two 20 minutes sessions per week with the elderly doing homework assigned by the activity group and log down the timing in the log book.This arrangement is to account for the placebo effect of additional social interaction time and attention that the treatment group will receive during this period.
  After completing the 1st 12 weeks' participation in the Waiting Control Group, the subject dyads in the waiting control group will receive the same training and treatment as the treatment group.
  Interventions: Other: acupressure

INTERVENTIONS:
Other: acupressure — A 15 minutes structured acupressure protocol with specific acupoints and applications technique will be performed on the elderly participants twice a week by the research team in YCHSS centers. The caregiver of the elderly will be trained and perform the same acupressure protocol on the elderly at 2 additional occasions during the week. The total trial period is 12 weeks.
  Other Names: Tui-na

SUMMARY:
Acupressure has been used for thousands of years in China. Through applying pressure on the specific acupoints based on TCM theory, acupressure could promote relaxation and wellness, balance yin-yang and treat diseases.

The PI has been using acupressure to treat various diseases in the clinics of the School of Chinese Medicine, HKU. Acupressure has demonstrated significant efficacy in treating geriatric diseases, obstetric diseases, pediatric diseases, rheumatoid arthritis and various painful symptoms. When applying acupressure on the Head- Neck - Shoulder area, it could also help to improve insomnia, reduce pain, and regulate the mood of the patients.

"Frailty" is a geriatric syndrome of growing importance in the medical field. Prevalence of frailty increases with age. As our life expectancy increase, there will be more elderly suffered from frailty in the later stage of their life. Although there is still a lack of universally accepted clinical definition for frailty, the syndrome is now commonly understood as decreased reserves in multiple systems, and lowered resilience to negative stress. Frailty could be initiated by single or multiple conditions including malnutrition, chronic diseases, lack of exercise, stress and physiological or social changes caused by aging. Its manifestation includes sarcopenia, anorexia, energy reduction, dysfunctional neuroendocrine system and a pro-inflammatory state. Frailty could affect the emotional state of the elderly, meanwhile, positive affect is protective against the functional and physical decline associated with frailty.[1] There is limited treatment or medication for frailty. The investigators believe that acupressure could be a possible non invasive means to improve the general health conditions, including the emotional conditions of the frail elderly. In the past 2 years, the school of Chinese Medicine has been promoting acupressure as a health maintenance technique to the elderly, mostly frail elderly living in the community dwelling through seminars. It is in our interest to run a prospective research to further understand the efficacy of acupressure in a wider range of frail elderly. The investigators would like to use a well-designed pragmatic randomized controlled trial (PRCT) to investigate if acupressure could help the frail elderly to improve their general quality of life.

DETAILED DESCRIPTION:
The research is a collaborative project by HKU and Yan Chai Hospital, with the aim of investigating the potential benefits of applying acupressure regularly on frail elderly. The study is designed as a prospective randomized control trial with the primary objective to investigate if acupressure could help the elderly to improve their general quality of life.

"Frailty" is a geriatric syndrome of growing importance in the medical field. Although there is still a lack of universally accepted clinical definition for frailty, the syndrome is now commonly understood as decreased reserves in multiple systems, and lowered resilience to negative stress. Frailty could affect the emotional state of the elderly; meanwhile, positive affect is protective against the functional and physical decline associated with frailty. Since there is limited treatment or medication for frailty. We would like to investigate if acupressure could be a possible non-invasive means to improve the general health conditions, including the psycho-social well being of the frail elderly.

The subjects of this study are the frail elderly living in the community dwellings who are members of the elderly centers. Our study is a pragmatic research comparing the acupressure treatment with care as usual, with the objectives of investigating

1. if a non invasive, easy to learn acupressure protocol could improve the general quality of life of the frail elderly
2. if there is a positive affect on the relationship between the informal caregiver and the elderly through practicing acupressure on the elderly by the caregiver

We will use the Tilburg Frail Indicator (TFI) as our frailty assessment instrument to identify the subjects for this study. The elderly will enroll with their informal caregiver as a dyad. Appropriate training (min 4 hours) and certification will be offered to the caregivers to ensure that they could practice the designed acupressure protocol on the elderly.

I. Trial Design This is a multicenter, pragmatic randomized control trial (PRCT) with a prospective design

Hypothesis:

Applying regular acupressure (4 times a week, totally 12 weeks) on frail elderly will improve one or more of the following aspects.

* Elderly's quality of life
* Elderly's psychological functioning
* Elderly's psychosocial functioning
* Elderly's sleeping quality
* Blood pressure/heart rate
* Caregiver's stress level

  140 frail elderlies currently served by the Social Centers for the elderly and Neighborhood Elderly Centers of the Yan Chai Hospital, Social Services Department (YCHSS) and their caregiver will be recruited. All accepted subjects will be in dyad, (i.e. 1 frail elderly and 1designated caregiver, who commits to learn and administered the acupressure procedure on the frail elderly according to the set protocol). All applications will be screened by the social worker in the centre based on the inclusion and exclusion criteria. Qualified applicants will be invited for a health assessment conducted by registered TCM practitioner in the research team to confirm their suitability and invite them to sign the consent form. The consented elderly-caregiver dyad will be allocated randomly into treatment group and waiting control group. Randomization is done by computer generated number list in block of 4.

II. Intervention Acupressure Group A 15 minutes structured acupressure protocol with specific acupoints and applications technique will be performed on the elderly participants twice a week by the research team in YCHSS centers. The caregiver of the elderly will be trained and perform the same acupressure protocol on the elderly at 2 additional occasions during the week. The total trial period is 12 weeks.

The acupressure treatment involved 12 steps, and mainly concentrates on the acupoints on face, head, neck and shoulder. The treatment is designed to be operated by layman. The acupoints chosen are all easy to be located. All the movements/steps selected are well established and commonly used in the TCM practices. Any movement that demand professional training or involve potential risk (e.g. joint mobilization) is excluded from the protocol. The total treatment process will last for approximately 15 mins.

Waiting Control group:

No acupressure therapy will be provided during the 1st 12 weeks' of study. The enrolled elderly will join a group activity, resembling the other group activities that held in that particular center, their caregivers will be requested to spend two 20 minutes sessions per week with the elderly doing homework assigned by the activity group and log down the timing in the LOG BOOK. This arrangement is to account for the placebo effect of additional social interaction time and attention that the treatment group will receive during this period. After completing the 1st 12 weeks' participation in the Waiting Control Group, the subject dyads in the waiting control group will receive the same training and treatment as the treatment group.

III. Measurement of efficacy and Data analysis Efficacy of the treatments will be measured in multi dimensions before and after the treatment for both groups. The measurement taken before the intervention will serve as the baseline, and the after treatment measurements will be taken (1) within 7days after the 12 weeks intervention and; (2) 3 months after the 12 weeks intervention completed. The primary outcomes will be the change in quality of life, psychological functioning, psychosocial functioning, sleeping quality and physiological aspects of the frail elderly. Secondary outcome will be the change of strain level of their caregivers. All instruments employed are international recognized and provide an absolute score in measurement.

ELIGIBILITY:
Inclusion Criteria:

* Elderly:

  1. Age: over 65 years old;
  2. Gender: male or female;
  3. Currently is a client served by the identified centers of YCHSS;
  4. Demonstrate frailty : score 5 or more in the Tilburg Frailty Indicator (TFI );
  5. Able to enroll in patient-caregiver dyad (i.e. have a capable designated caregiver enroll in the trial). The caregiver is preferred to be a family member, but could also be a close friend or helper, as long as the designated person spends time regularly with the frail elderly;
  6. Physically fit to sit on a normal chair for 15-20 mins for acupressure treatment;
  7. Cognitively competent to understand the instruction from the practitioner and participate actively in the control group activity (resembling other art and craft activities offered by center);
  8. Cognitively competent to sign the consent form: score 6 or more in Abbreviated Mental Test (AMT, Hong Kong Version);
  9. Signed the Patient/Subject Consent Form for this study.

Caregiver:

1. Family member, paid/informal helper or friend of the qualified elderly who will meet with the elderly on a weekly basis;
2. Committed to learn the acupressure protocol and practice the protocol on the elderly twice a week, during the 12-weeks study period, and support the control group activities (if applicable);
3. Cognitively competent to sign the consent form (for caregiver age 65 or above): score 6 or more in Abbreviated Mental Test (AMT, Hong Kong Version,);
4. Signed the Patient/Subject Consent Form for this study.

Exclusion Criteria:

* Elderly in the following situation will be excluded from the study:

  1. Who is currently receiving acupressure as a regular therapy;
  2. Who is decision impaired and unfit to sign the consent form;
  3. Who is suffering from one of the related contraindications for acupressure ( including open sores; undiagnosed rashes; high fever; hypertensive emergence; sore and enlarged lymph nodes; the site of an injury, surgery or injection; burn wounds; skin ulcers and eczema);
  4. Who is unable to comply to the set treatment schedule (20% non compliance is allowed).

Caregiver in the following situation will be excluded from the study:

1. Who do not complete the training or incapable to reach a set standard of performing the acupressure protocol;
2. Who is decision impaired and unfit to sign the consent form.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 106 (Actual)
Dates: Start 2014-12; Primary Completion 2015-10 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Elderlies' Quality of Life | Time Frame: Baseline, change from baseline at 3rd month, change from baseline at 6th month
  Questionnaires:
  1. General QOL: WHOQOL-BREF, Interview Version for Hong Kong Chinese(28 Items)[2]
  2. Psychosocial function: Geriatric Depression Scale SF(15 Items)[4]
  3. Sleeping quality: PSQI(9 Items)[5]
  Physiological aspect: Electronic sphygmomanometer:Blood pressure and Heart rate

SECONDARY OUTCOMES:
Caregiver Stress Level Modified Care givers Strain Index(13 items)[6]; Perceived burden level scale （1 item） | Time Frame: Baseline, change from baseline at 3rd month, change from baseline at 6th month
  Questionnaire:
  Modified Care givers Strain Index(13 items)[6]; Perceived burden level scale （1 item）.

CONTACTS AND LOCATIONS:
Overall Officials: Lei Li, Principal Investigator — The University of Hong Kong
Locations (1):
- School of Chinese Medicine, The University of Hong Kong, Hong Kong, Hong Kong, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Ostir GV, Ottenbacher KJ, Markides KS. Onset of frailty in older adults and the protective role of positive affect. Psychol Aging. 2004 Sep;19(3):402-8. doi: 10.1037/0882-7974.19.3.402. PMID 15382991
- [Background] Hankins M. The reliability of the twelve-item general health questionnaire (GHQ-12) under realistic assumptions. BMC Public Health. 2008 Oct 14;8:355. doi: 10.1186/1471-2458-8-355. PMID 18854015
- [Background] SHEIKH JI, YESAVAGE JA. Geriatric Depression Scale (GDS): recent evidence and development of a shorter version. Clin Gerontol . 1986 June;5(1/2):165-173.
- [Background] Buysse DJ, Reynolds CF 3rd, Monk TH, Berman SR, Kupfer DJ. The Pittsburgh Sleep Quality Index: a new instrument for psychiatric practice and research. Psychiatry Res. 1989 May;28(2):193-213. doi: 10.1016/0165-1781(89)90047-4. PMID 2748771